CLINICAL TRIAL: NCT02692963
Title: Safety and Protective Efficacy of BCG Vaccination Against Controlled Human Malaria Infection
Acronym: BCG-EHMI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: BCG-EHMI; 2015-005735-40 (EudraCT Number); NL56222.091.15 (Other: Central Committee on Research Involving Human Subjects (CCMO) of The Netherlands)
Record Dates: First submitted 2016-02-02; First posted 2016-02-26 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2016-08

CONDITIONS: Malaria; Plasmodium Falciparum
MeSH Terms: conditions — Malaria; Malaria, Falciparum

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BCG vaccination (Experimental)
  Interventions: Biological: BCG vaccination
- Control (No Intervention)

INTERVENTIONS:
Biological: BCG vaccination — BCG vaccine InterVax
  Arms: BCG vaccination

SUMMARY:
The Bacillus Calmette-Guérin (BCG) vaccine, a live attenuated Mycobacterium bovis vaccine, has been used to prevent tuberculosis for almost a century, and it is still the most used vaccine in the world. There is also circumstantial and indirect evidence that BCG vaccination can protect against malaria. Investigators hypothesize that BCG vaccination can offer protection against malaria in the Controlled Human Malaria Infection (CHMI) model.

A total of 20 healthy male and female volunteers will participate in this randomized, single-blind clinical trial. Volunteers will be randomized to receive either BCG vaccination (BCG vaccine SSI) (group 1, n=10) or no treatment (group 2, n=10). Five weeks after vaccination of group 1 volunteers, all volunteers will undergo a CHMI administered by the bites of five P. falciparum infected Anopheles mosquitoes.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is aged ≥18 and ≤35 years and in good health.
2. Subject has adequate understanding of the procedures of the study and agrees to abide strictly thereby.
3. Subject is able to communicate well with the investigator and is available to attend all study visits.
4. The subject will remain within the Netherlands during the challenge period, not travel to a malaria-endemic area during the study period, and is reachable (24/7) by mobile telephone throughout the entire study period.
5. Subject agrees to inform his/her general practitioner about participation in the study and to sign a request to release by the General Practitioner (GP), and medical specialist when necessary, any relevant medical information concerning possible contra-indications for participation in the study.
6. The subject agrees to refrain from blood donation to Sanquin or for other purposes throughout the study period and for a defined period thereafter according to current Sanquin guidelines.
7. For female subjects: subject agrees to use adequate contraception and not to breastfeed for the duration of study.
8. Subject agrees to refrain from intensive physical exercise (disproportionate to the subjects usual daily activity or exercise routine) during the malaria challenge period.
9. Subject has signed informed consent.

Exclusion Criteria:

1. Any history, or evidence at screening, of clinically significant symptoms, physical signs or abnormal laboratory values suggestive of systemic conditions, such as cardiovascular, pulmonary, renal, hepatic, neurological, dermatological, endocrine, malignant, haematological, infectious, immunodeficient, psychiatric and other disorders, which could compromise the health of the volunteer during the study or interfere with the interpretation of the study results. These include, but are not limited to, any of the following.

   1.1 Body weight <50 kg or Body Mass lndex (BM l) <18 or >30 kg/m2 at screening. 1.2 A heightened risk of cardiovascular disease, as determined by: an estimated ten year risk of fatal cardiovascular disease of >5% at screening, as determined by the Systematic Coronary Risk Evaluation (SCORE); history, or evidence at screening, of clinically significant arrhythmia's, prolonged QT-interval or other clinically relevant ECG abnormalities; or a positive family history of cardiac events in 1st or 2nd degree relatives <50 years old.

   1.3 A medical history of functional asplenia, sickle cell trait disease, thalassaemia trait/disease or G6PD deficiency.

   1.4 History of epilepsy in the period of five years prior to study onset, even if no longer on medication.

   1.5 Screening tests positive for Human immunodeficiency Virus (HlV), or active Hepatitis B Virus (HBS) or Hepatitis C Virus (HCV).

   1.6 Chronic use of i) immunosuppressive drugs, ii) antibiotics, iii) or other immune modifying drugs within three months prior to study onset (inhaled and topical corticosteroids and oral anti-histamines exempted) or expected use of such during the study period.

   1.7 Use of Non-steroidal Anti-inflammatory Drugs (NSAlDs) in the four weeks prior to study start or expected use of NSAIDS during the study period.

   1.8 History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years.

   1.9 Any history of treatment for severe psychiatric disease by a psychiatrist in the past year.

   1.10 History of drug or alcohol abuse interfering with normal social function in the period of one year prior to study onset, positive urine toxicology test for cocaine or amphetamines at screening or prior to infection, or positive urine toxicology test for cannabis at inclusion.
2. For female subjects: positive urine pregnancy test at screening or at inclusion.
3. Any history of malaria, positive serology for P. falciparum, or previous participation in any malaria (vaccine) study.
4. Known hypersensitivity to or contra-indications (including co-medication) for use of chloroquine, Malarone or artemether-lumefantrine, or history of severe (allergic) reactions to mosquito bites.
5. Receipt of any vaccinations in the 3 months prior to the start of the study or plans to receive any other vaccinations during the study period or up to 90 days thereafter.
6. Participation in any other clinical study in the 30 days prior to the start of the study or during the study period.
7. Being an employee or student of the department of Medical Microbiology of the Radboudumc or the department of lnternal Medicine.
8. Previous BCG-vaccination; history of tuberculosis or positive Mantoux test; or positive whole blood interferon-gamma (IFN-γ) response to restimulation with M. tuberculosis at screening.
9. Any other condition or situation that would, in the opinion of the investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-04; Primary Completion 2016-10 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Frequency and magnitude of adverse events | day of BCG vaccination until day 37 after malaria challenge infection
  Adverse event collection and routine safety and hematology laboratory evaluations will be conducted from the day of BCG vaccination until day 37 after CHMI.
Time to blood stage parasitemia detectable by qPCR | day 1 - 21 after malaria challenge infection
  The effectiveness of BCG vaccination to protect against CHMI will be evaluated by quantitative PCR.

SECONDARY OUTCOMES:
Changes in cellular (innate and adaptive) immune responses | inclusion until day 120 after malaria challenge infection
Changes in plasma cytokine levels | inclusion until day 120 after malaria challenge infection

CONTACTS AND LOCATIONS:
Overall Officials: Robert Sauerwein, Prof., Principal Investigator — Radboud University Medical Center; Mihai Netea, Prof., Principal Investigator — Radboud University Medical Center; Jona Walk, MD, Study Director — Radboud University Medical Center
Locations (1):
- Radboud university medical center, Nijmegen, Netherlands